CLINICAL TRIAL: NCT02692144
Title: Effect of an Optimized Savory Cluster on Glycemic and Insulinemic Responses in Healthy Individuals: A Randomized, Cross-over Study
Brief Title: Effect of an Optimized Savory Cluster on Glycemic and Insulinemic Responses in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1511
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Peak Rise of Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test-cluster (Experimental): 56g of optimized savory cluster made through a proprietary process with slowly digestible carbohydrates and fiber
  Interventions: Other: Test Cluster
- Control-cluster (Placebo Comparator): 56g of control cluster made from general baking process with typical ingredients commonly used in commercially available energy snacks or bars
  Interventions: Other: Test Cluster
- White-bread (Placebo Comparator): 47g of white bread containing equivalent amount of available carbohydrate in 56g of optimized savory cluster
  Interventions: Other: Test Cluster

INTERVENTIONS:
Other: Test Cluster — Test cluster is an optimized savory cluster made through a proprietary baking process combined with slow digestible carbohydrates and fiber

SUMMARY:
This study was to test the hypothesis that an optimized savory cluster (Test-cluster) made through a proprietary baking process combined with slow digestible carbohydrates and fiber will elicit lower postprandial blood glucose and insulin responses than a Control-cluster made from general processing procedure and with typical ingredients commonly used in commercially available snacks or bars: oats, peanuts, and corn syrup. However, since the Test-cluster contains ~30% less available-carbohydrate (24g) than the Control (33g), the postprandial responses elicited by the Test-cluster was also compared with those after a portion of White-bread matched for available-carbohydrate content. On 3 separate days, 25 healthy male or non-pregnant females aged 18-60 yr with BMI between 20 and 35 kg/m² with fasting serum glucose <7.0mmol/L (126 mg/dL) were asked to consume 1 serving (56g) of the Test- or Control-cluster or 47g White Bread and had blood glucose and insulin measured at intervals over the next 4 hr. Each serving of Test-cluster and Control-cluster contained similar amounts of total carbohydrates, protein, fat and energy content. Each serving of Test-cluster and White-bread had equivalent amount of 24g available carbohydrate.

On each test occasion, after subjects were weighed, 2 fasting blood samples were obtained by finger-prick 5min apart and after the 2nd sample, the subject started to consume a test meal. Subjects were asked to consume the entire test meal within 10 min. At the first bite a timer was started and blood samples for were taken for glucose analysis at 10, 20, 30, 40, 50, 60, 90, 120, 180 and 240 min after starting to eat. Additional blood was taken into a separate vial at -5, 0, 20, 40, 60, 90, 120, 180 and 240 min for insulin analysis. Blood samples were obtained from hands warmed with an electric heating pad for 3-5 min prior to each sample. During the 4hr of the test, participants remained seated quietly. After the last blood sample participants were offered a snack and then allowed to leave.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females, 18-60 years of age, inclusive
* Body mass index (BMI) ≥ 20.0 and < 35 kg/m² at screening (visit 1).
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
* Normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Peak rise of blood glucose | 0-4 hours post consumption

SECONDARY OUTCOMES:
Incremental area under the curve of blood glucose | 0-4 hours post consumption
Peak rise of serum insulin | 0-4 hours post consumption
Incremental area under the curve of serum insulin | 0-4 hours post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, PhD, Principal Investigator — GI Laboratories

IPD SHARING:
Plan to Share IPD: No